CLINICAL TRIAL: NCT00355316
Title: Peripheral Blood Molecular Staging of Breast Cancer: A Prospective Cohort Study Designed to Determine the Clinical Significance of Molecular Detection of Breast Cancer in the Peripheral Blood of Stage IV Breast Cancer Patients
Brief Title: A Study to Determine the Clinical Significance of Molecular Detection of Breast Cancer in the Blood of Stage IV Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 05-0435 / 201109033
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Peripheral; Blood
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stage IV Breast Cancer (Experimental): Blood draws at baseline before systemic therapy. Blood draw then every 6 weeks for approximately 12 weeks.
  Interventions: Other: Blood draw
- Healthy Volunteers (Other): Baseline blood draw.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw

SUMMARY:
This study is designed to determine whether molecular detection of breast cancer cells in the peripheral blood of Stage IV breast cancer patients is a clinically relevant predictor of progression-free and overall survival. Stage IV breast cancer patients who have measurable breast cancer metastases and are initiating a regimen of systemic therapy are eligible for enrollment. Multi-marker real-time RT-PCR analysis will be performed on peripheral blood specimens from 92 breast cancer patients and 120 healthy volunteers. Peripheral blood specimens from breast cancer patients will be obtained at the time of study entry (prior to initiation of systemic therapy) and at serial time points during follow-up. Subjects will be followed longitudinally until death, although the study has been powered so that the primary objective can be addressed after 12 months of follow-up. Healthy volunteers will be asked to provide a blood sample at time of enrollment but will not be followed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - Stage IV breast cancer patients

1. Patient age must be > 21 years.
2. Patient must have a tissue diagnosis of invasive breast cancer.
3. Patient must have documented evidence of metastatic disease.
4. Patient must have measurable lesions.
5. Patients must be initiating systemic therapy. Patients receiving hormonal therapy, and/or chemotherapy alone or in combination with other therapies are eligible.
6. Patient must have an ECOG performance status of 0, 1, or 2.
7. Patient must be available for follow-up.
8. Patient or their authorized legally acceptable representative must consent to be in the study and must have signed and dated an approved consent form which conforms to federal and institutional guidelines.
9. The patient with a previous history of non-breast malignancy is eligible for this study only if the patient meets the following criteria for a cancer survivor. A cancer survivor is eligible provided the following criteria are met: (1) patient has undergone potentially curative therapy for all prior malignancies, (2) patients have been considered disease free for at least 5 years (with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix).

Inclusion Criteria - Healthy volunteers

A volunteer will be eligible for inclusion in this study only if ALL of the following criteria apply:

1. Volunteer age must be > 21 years.
2. Volunteer or their authorized legally acceptable representative must consent to be in the study and must have signed and dated an approved consent form which conforms to federal and institutional guidelines.
3. Patients with benign breast disease are eligible for enrollment.
4. The volunteer with a previous history of non-breast malignancy is eligible for this study only if the patient meets the following criteria for a cancer survivor. A cancer survivor is eligible provided both of the following criteria are met: (1) patient has undergone potentially curative therapy for all prior malignancies, (2) patient has been considered disease free for at least 5 years (with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix).

Exclusion Criteria:

Exclusion Criteria - Stage IV breast cancer patients

A patient will be ineligible for inclusion in this study if ANY of the following criteria apply:

1. No documented metastatic disease.
2. No measurable lesions.
3. Bone only and/or brain metastasis.
4. Patient is not initiating a new regimen of systemic therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2005-11; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The prevalence of breast cancer cells in the peripheral blood | 1 year
  Specifically, it is predicted that 60% of subjects with Stage IV breast cancer will have evidence of breast cancer cells in the peripheral blood by multi-marker real-time RT-PCR analysis, and that these subjects will experience a significantly decreased progression-free and overall survival.

SECONDARY OUTCOMES:
Evaluate the prognostic significance of molecular detection of breast cancer cells in peripheral blood after initiation of systemic therapy. | Until patient death
  Specifically, we will determine if molecular detection of circulating breast cancer cells after the initiation of systemic therapy is associated with a significantly decreased progression-free and overall survival.
Quantify baseline molecular marker expression levels in the peripheral blood of healthy volunteers | Approximately 12 weeks
  Determine if baseline molecular marker expression levels are dependent on patient age, race, and/or the presence of benign breast disease.
Compare molecular analyses to the results of the CellSeach assay | Approximately 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William E. Gillanders, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Background] Valagussa P, Bonadonna G, Veronesi U. Patterns of relapse and survival following radical mastectomy. Analysis of 716 consecutive patients. Cancer. 1978 Mar;41(3):1170-8. doi: 10.1002/1097-0142(197803)41:33.0.co;2-i. PMID 638961
- [Background] Ghossein RA, Carusone L, Bhattacharya S. Review: polymerase chain reaction detection of micrometastases and circulating tumor cells: application to melanoma, prostate, and thyroid carcinomas. Diagn Mol Pathol. 1999 Dec;8(4):165-75. doi: 10.1097/00019606-199912000-00001. PMID 10617272
- [Background] Diel IJ, Kaufmann M, Goerner R, Costa SD, Kaul S, Bastert G. Detection of tumor cells in bone marrow of patients with primary breast cancer: a prognostic factor for distant metastasis. J Clin Oncol. 1992 Oct;10(10):1534-9. doi: 10.1200/JCO.1992.10.10.1534. PMID 1403032
- [Background] Allard WJ, Matera J, Miller MC, Repollet M, Connelly MC, Rao C, Tibbe AG, Uhr JW, Terstappen LW. Tumor cells circulate in the peripheral blood of all major carcinomas but not in healthy subjects or patients with nonmalignant diseases. Clin Cancer Res. 2004 Oct 15;10(20):6897-904. doi: 10.1158/1078-0432.CCR-04-0378. PMID 15501967
- [Background] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Background] Baker MK, Mikhitarian K, Osta W, Callahan K, Hoda R, Brescia F, Kneuper-Hall R, Mitas M, Cole DJ, Gillanders WE. Molecular detection of breast cancer cells in the peripheral blood of advanced-stage breast cancer patients using multimarker real-time reverse transcription-polymerase chain reaction and a novel porous barrier density gradient centrifugation technology. Clin Cancer Res. 2003 Oct 15;9(13):4865-71. PMID 14581359
- [Background] Berns EM, Klijn JG, van Putten WL, van Staveren IL, Portengen H, Foekens JA. c-myc amplification is a better prognostic factor than HER2/neu amplification in primary breast cancer. Cancer Res. 1992 Mar 1;52(5):1107-13. PMID 1737370
- [Background] Datta YH, Adams PT, Drobyski WR, Ethier SP, Terry VH, Roth MS. Sensitive detection of occult breast cancer by the reverse-transcriptase polymerase chain reaction. J Clin Oncol. 1994 Mar;12(3):475-82. doi: 10.1200/JCO.1994.12.3.475. PMID 7509852
- [Background] Gasparini G, Toi M, Gion M, Verderio P, Dittadi R, Hanatani M, Matsubara I, Vinante O, Bonoldi E, Boracchi P, Gatti C, Suzuki H, Tominaga T. Prognostic significance of vascular endothelial growth factor protein in node-negative breast carcinoma. J Natl Cancer Inst. 1997 Jan 15;89(2):139-47. doi: 10.1093/jnci/89.2.139. PMID 8998183
- [Background] Ioachim E, Kamina S, Athanassiadou S, Agnantis NJ. The prognostic significance of epidermal growth factor receptor (EGFR), C-erbB-2, Ki-67 and PCNA expression in breast cancer. Anticancer Res. 1996 Sep-Oct;16(5B):3141-7. PMID 8920782
- [Background] Anan K, Morisaki T, Katano M, Ikubo A, Tsukahara Y, Kojima M, Uchiyama A, Kuroki S, Torisu M, Tanaka M. Assessment of c-erbB2 and vascular endothelial growth factor mRNA expression in fine-needle aspirates from early breast carcinomas: pre-operative determination of malignant potential. Eur J Surg Oncol. 1998 Feb;24(1):28-33. doi: 10.1016/s0748-7983(98)80121-2. PMID 9542512
- [Background] Bieche I, Lazar V, Nogues C, Poynard T, Giovangrandi Y, Bellet D, Lidereau R, Vidaud M. Prognostic value of chorionic gonadotropin beta gene transcripts in human breast carcinoma. Clin Cancer Res. 1998 Mar;4(3):671-6. PMID 9533536
- [Background] Harbeck N, Dettmar P, Thomssen C, Henselmann B, Kuhn W, Ulm K, Janicke F, Hofler H, Graeff H, Schmitt M. Prognostic impact of tumor biological factors on survival in node-negative breast cancer. Anticancer Res. 1998 May-Jun;18(3C):2187-97. PMID 9703782
- [Background] Linderholm B, Tavelin B, Grankvist K, Henriksson R. Vascular endothelial growth factor is of high prognostic value in node-negative breast carcinoma. J Clin Oncol. 1998 Sep;16(9):3121-8. doi: 10.1200/JCO.1998.16.9.3121. PMID 9738584
- [Background] Lockett MA, Baron PL, O'Brien PH, Elliott BM, Robison JG, Maitre N, Metcalf JS, Cole DJ. Detection of occult breast cancer micrometastases in axillary lymph nodes using a multimarker reverse transcriptase-polymerase chain reaction panel. J Am Coll Surg. 1998 Jul;187(1):9-16. doi: 10.1016/s1072-7515(98)00130-6. PMID 9660019
- [Background] Lockett MA, Metcalf JS, Baron PL, O'Brien PH, Elliott BM, Robison JG, Cole DJ. Efficacy of reverse transcriptase-polymerase chain reaction screening for micrometastic disease in axillary lymph nodes of breast cancer patients. Am Surg. 1998 Jun;64(6):539-43; discussion 543-4. PMID 9619175
- [Background] Molina R, Jo J, Filella X, Zanon G, Pahisa J, Mu noz M, Farrus B, Latre ML, Escriche C, Estape J, Ballesta AM. c-erbB-2 oncoprotein, CEA, and CA 15.3 in patients with breast cancer: prognostic value. Breast Cancer Res Treat. 1998 Sep;51(2):109-19. doi: 10.1023/a:1005734429304. PMID 9879773
- [Background] Pathak KA, Khanna R, Khanna HD, Khanna S, Gupta S, Khanna NN. Carcinoembryonic antigen: an invaluable marker for advanced breast cancer. J Postgrad Med. 1996 Jul-Sep;42(3):68-71. PMID 9715319
- [Background] Mitas M, Mikhitarian K, Walters C, Baron PL, Elliott BM, Brothers TE, Robison JG, Metcalf JS, Palesch YY, Zhang Z, Gillanders WE, Cole DJ. Quantitative real-time RT-PCR detection of breast cancer micrometastasis using a multigene marker panel. Int J Cancer. 2001 Jul 15;93(2):162-71. doi: 10.1002/ijc.1312. PMID 11410861
- [Background] Gillanders WE, Mikhitarian K, Hebert R, Mauldin PD, Palesch Y, Walters C, Urist MM, Mann GB, Doherty G, Herrmann VM, Hill AD, Eremin O, El-Sheemy M, Orr RK, Valle AA, Henderson MA, Dewitty RL, Sugg SL, Frykberg E, Yeh K, Bell RM, Metcalf JS, Elliott BM, Brothers T, Robison J, Mitas M, Cole DJ. Molecular detection of micrometastatic breast cancer in histopathology-negative axillary lymph nodes correlates with traditional predictors of prognosis: an interim analysis of a prospective multi-institutional cohort study. Ann Surg. 2004 Jun;239(6):828-37; discussion 837-40. doi: 10.1097/01.sla.0000128687.59439.d6. PMID 15166962
- [Background] Mitas M, Hoover L, Silvestri G, Reed C, Green M, Turrisi AT, Sherman C, Mikhitarian K, Cole DJ, Block MI, Gillanders WE. Lunx is a superior molecular marker for detection of non-small cell lung cancer in peripheral blood [corrected]. J Mol Diagn. 2003 Nov;5(4):237-42. doi: 10.1016/s1525-1578(10)60480-1. PMID 14573783
- [Background] Campana D, Pui CH. Detection of minimal residual disease in acute leukemia: methodologic advances and clinical significance. Blood. 1995 Mar 15;85(6):1416-34. No abstract available. PMID 7888664
- [Background] Cave H, Guidal C, Rohrlich P, Delfau MH, Broyart A, Lescoeur B, Rahimy C, Fenneteau O, Monplaisir N, d'Auriol L, et al. Prospective monitoring and quantitation of residual blasts in childhood acute lymphoblastic leukemia by polymerase chain reaction study of delta and gamma T-cell receptor genes. Blood. 1994 Apr 1;83(7):1892-902. PMID 8142656
- [Background] Roberts WM, Estrov Z, Ouspenskaia MV, Johnston DA, McClain KL, Zipf TF. Measurement of residual leukemia during remission in childhood acute lymphoblastic leukemia. N Engl J Med. 1997 Jan 30;336(5):317-23. doi: 10.1056/NEJM199701303360501. PMID 9011783
- [Background] Pallisgaard N, Clausen N, Schroder H, Hokland P. Rapid and sensitive minimal residual disease detection in acute leukemia by quantitative real-time RT-PCR exemplified by t(12;21) TEL-AML1 fusion transcript. Genes Chromosomes Cancer. 1999 Dec;26(4):355-65. doi: 10.1002/(sici)1098-2264(199912)26:43.0.co;2-3. PMID 10534771
- [Background] Mensink E, van de Locht A, Schattenberg A, Linders E, Schaap N, Geurts van Kessel A, De Witte T. Quantitation of minimal residual disease in Philadelphia chromosome positive chronic myeloid leukaemia patients using real-time quantitative RT-PCR. Br J Haematol. 1998 Aug;102(3):768-74. doi: 10.1046/j.1365-2141.1998.00823.x. PMID 9722305
- [Background] Nakao M, Janssen JW, Flohr T, Bartram CR. Rapid and reliable quantification of minimal residual disease in acute lymphoblastic leukemia using rearranged immunoglobulin and T-cell receptor loci by LightCycler technology. Cancer Res. 2000 Jun 15;60(12):3281-9. PMID 10866322
- [Background] Emig M, Saussele S, Wittor H, Weisser A, Reiter A, Willer A, Berger U, Hehlmann R, Cross NC, Hochhaus A. Accurate and rapid analysis of residual disease in patients with CML using specific fluorescent hybridization probes for real time quantitative RT-PCR. Leukemia. 1999 Nov;13(11):1825-32. doi: 10.1038/sj.leu.2401566. PMID 10557058
- [Background] Cassinat B, Zassadowski F, Balitrand N, Barbey C, Rain JD, Fenaux P, Degos L, Vidaud M, Chomienne C. Quantitation of minimal residual disease in acute promyelocytic leukemia patients with t(15;17) translocation using real-time RT-PCR. Leukemia. 2000 Feb;14(2):324-8. doi: 10.1038/sj.leu.2401652. PMID 10673752
- [Background] Stathopoulou A, Vlachonikolis I, Mavroudis D, Perraki M, Kouroussis Ch, Apostolaki S, Malamos N, Kakolyris S, Kotsakis A, Xenidis N, Reppa D, Georgoulias V. Molecular detection of cytokeratin-19-positive cells in the peripheral blood of patients with operable breast cancer: evaluation of their prognostic significance. J Clin Oncol. 2002 Aug 15;20(16):3404-12. doi: 10.1200/JCO.2002.08.135. PMID 12177100
- [Background] Gradilone A, Gazzaniga P, Silvestri I, Gandini O, Trasatti L, Lauro S, Frati L, Agliano AM. Detection of CK19, CK20 and EGFR mRNAs in peripheral blood of carcinoma patients: correlation with clinical stage of disease. Oncol Rep. 2003 Jan-Feb;10(1):217-22. PMID 12469172
- [Background] Galan M, Vinolas N, Colomer D, Soler G, Munoz M, Longaron R, Ventura PJ, Gascon P, Estape J. Detection of occult breast cancer cells by amplification of CK19 mRNA by reverse transcriptase-polymerase chain reaction: role of surgical manipulation. Anticancer Res. 2002 Sep-Oct;22(5):2877-84. PMID 12530011
- [Background] Xenidis N, Vlachonikolis I, Mavroudis D, Perraki M, Stathopoulou A, Malamos N, Kouroussis C, Kakolyris S, Apostolaki S, Vardakis N, Lianidou E, Georgoulias V. Peripheral blood circulating cytokeratin-19 mRNA-positive cells after the completion of adjuvant chemotherapy in patients with operable breast cancer. Ann Oncol. 2003 Jun;14(6):849-55. doi: 10.1093/annonc/mdg259. PMID 12796021
- [Background] Weigelt B, Bosma AJ, Hart AA, Rodenhuis S, van 't Veer LJ. Marker genes for circulating tumour cells predict survival in metastasized breast cancer patients. Br J Cancer. 2003 Apr 7;88(7):1091-4. doi: 10.1038/sj.bjc.6600868. PMID 12671691
- [Background] Zach O, Kasparu H, Krieger O, Hehenwarter W, Girschikofsky M, Lutz D. Detection of circulating mammary carcinoma cells in the peripheral blood of breast cancer patients via a nested reverse transcriptase polymerase chain reaction assay for mammaglobin mRNA. J Clin Oncol. 1999 Jul;17(7):2015-9. doi: 10.1200/JCO.1999.17.7.2015. PMID 10561252
- [Background] Bossolasco P, Ricci C, Farina G, Soligo D, Pedretti D, Scanni A, Deliliers GL. Detection of micrometastatic cells in breast cancer by RT-pCR for the mammaglobin gene. Cancer Detect Prev. 2002;26(1):60-3. doi: 10.1016/s0361-090x(02)00009-0. PMID 12088204
- [Background] Lin YC, Wu Chou YH, Liao IC, Cheng AJ. The expression of mammaglobin mRNA in peripheral blood of metastatic breast cancer patients as an adjunct to serum tumor markers. Cancer Lett. 2003 Feb 28;191(1):93-9. doi: 10.1016/s0304-3835(02)00545-1. PMID 12609714
- [Background] Zippelius A, Kufer P, Honold G, Kollermann MW, Oberneder R, Schlimok G, Riethmuller G, Pantel K. Limitations of reverse-transcriptase polymerase chain reaction analyses for detection of micrometastatic epithelial cancer cells in bone marrow. J Clin Oncol. 1997 Jul;15(7):2701-8. doi: 10.1200/JCO.1997.15.7.2701. PMID 9215843
- [Background] von Knebel Doeberitz M, Lacroix J. Nucleic acid based techniques for the detection of rare cancer cells in clinical samples. Cancer Metastasis Rev. 1999;18(1):43-64. doi: 10.1023/a:1006208303075. PMID 10505545
- [Background] Pantel K, Cote RJ, Fodstad O. Detection and clinical importance of micrometastatic disease. J Natl Cancer Inst. 1999 Jul 7;91(13):1113-24. doi: 10.1093/jnci/91.13.1113. PMID 10393719
- [Background] Salerno CT, Frizelle S, Niehans GA, Ho SB, Jakkula M, Kratzke RA, Maddaus MA. Detection of occult micrometastases in non-small cell lung carcinoma by reverse transcriptase-polymerase chain reaction. Chest. 1998 Jun;113(6):1526-32. doi: 10.1378/chest.113.6.1526. PMID 9631789
- [Background] Castaldo G, Tomaiuolo R, Sanduzzi A, Bocchino ML, Ponticiello A, Barra E, Vitale D, Bariffi F, Sacchetti L, Salvatore F. Lung cancer metastatic cells detected in blood by reverse transcriptase-polymerase chain reaction and dot-blot analysis. J Clin Oncol. 1997 Nov;15(11):3388-93. doi: 10.1200/JCO.1997.15.11.3388. PMID 9363870
- [Background] Dingemans AM, Brakenhoff RH, Postmus PE, Giaccone G. Detection of cytokeratin-19 transcripts by reverse transcriptase-polymerase chain reaction in lung cancer cell lines and blood of lung cancer patients. Lab Invest. 1997 Sep;77(3):213-20. PMID 9314945
- [Background] Jung R, Kruger W, Hosch S, Holweg M, Kroger N, Gutensohn K, Wagener C, Neumaier M, Zander AR. Specificity of reverse transcriptase polymerase chain reaction assays designed for the detection of circulating cancer cells is influenced by cytokines in vivo and in vitro. Br J Cancer. 1998 Nov;78(9):1194-8. doi: 10.1038/bjc.1998.653. PMID 9820179
- [Background] Bostick PJ, Chatterjee S, Chi DD, Huynh KT, Giuliano AE, Cote R, Hoon DS. Limitations of specific reverse-transcriptase polymerase chain reaction markers in the detection of metastases in the lymph nodes and blood of breast cancer patients. J Clin Oncol. 1998 Aug;16(8):2632-40. doi: 10.1200/JCO.1998.16.8.2632. PMID 9704713
- [Background] Martell M, Gomez J, Esteban JI, Sauleda S, Quer J, Cabot B, Esteban R, Guardia J. High-throughput real-time reverse transcription-PCR quantitation of hepatitis C virus RNA. J Clin Microbiol. 1999 Feb;37(2):327-32. doi: 10.1128/JCM.37.2.327-332.1999. PMID 9889212
- [Background] Bieche I, Olivi M, Champeme MH, Vidaud D, Lidereau R, Vidaud M. Novel approach to quantitative polymerase chain reaction using real-time detection: application to the detection of gene amplification in breast cancer. Int J Cancer. 1998 Nov 23;78(5):661-6. doi: 10.1002/(sici)1097-0215(19981123)78:53.0.co;2-i. PMID 9808539
- [Background] Hardingham JE, Kotasek D, Farmer B, Butler RN, Mi JX, Sage RE, Dobrovic A. Immunobead-PCR: a technique for the detection of circulating tumor cells using immunomagnetic beads and the polymerase chain reaction. Cancer Res. 1993 Aug 1;53(15):3455-8. PMID 8101760
- [Background] Denis MG, Lipart C, Leborgne J, LeHur PA, Galmiche JP, Denis M, Ruud E, Truchaud A, Lustenberger P. Detection of disseminated tumor cells in peripheral blood of colorectal cancer patients. Int J Cancer. 1997 Oct 21;74(5):540-4. doi: 10.1002/(sici)1097-0215(19971021)74:53.0.co;2-a. PMID 9355978
- [Background] Naume B, Borgen E, Beiske K, Herstad TK, Ravnas G, Renolen A, Trachsel S, Thrane-Steen K, Funderud S, Kvalheim G. Immunomagnetic techniques for the enrichment and detection of isolated breast carcinoma cells in bone marrow and peripheral blood. J Hematother. 1997 Apr;6(2):103-14. doi: 10.1089/scd.1.1997.6.103. PMID 9131439
- [Background] Eaton MC, Hardingham JE, Kotasek D, Dobrovic A. Immunobead RT-PCR: a sensitive method for detection of circulating tumor cells. Biotechniques. 1997 Jan;22(1):100-5. doi: 10.2144/97221st01. PMID 8994656
- [Background] Soria JC, Gauthier LR, Raymond E, Granotier C, Morat L, Armand JP, Boussin FD, Sabatier L. Molecular detection of telomerase-positive circulating epithelial cells in metastatic breast cancer patients. Clin Cancer Res. 1999 May;5(5):971-5. PMID 10353728
- [Background] Zhong XY, Kaul S, Lin YS, Eichler A, Bastert G. Sensitive detection of micrometastases in bone marrow from patients with breast cancer using immunomagnetic isolation of tumor cells in combination with reverse transcriptase/polymerase chain reaction for cytokeratin-19. J Cancer Res Clin Oncol. 2000 Apr;126(4):212-8. doi: 10.1007/s004320050035. PMID 10782894
- [Background] Rosenberg R, Gertler R, Friederichs J, Fuehrer K, Dahm M, Phelps R, Thorban S, Nekarda H, Siewert JR. Comparison of two density gradient centrifugation systems for the enrichment of disseminated tumor cells in blood. Cytometry. 2002 Dec 1;49(4):150-8. doi: 10.1002/cyto.10161. PMID 12454978
- [Background] Mitas M, Cole DJ, Hoover L, Fraig MM, Mikhitarian K, Block MI, Hoffman BJ, Hawes RH, Gillanders WE, Wallace MB. Real-time reverse transcription-PCR detects KS1/4 mRNA in mediastinal lymph nodes from patients with non-small cell lung cancer. Clin Chem. 2003 Feb;49(2):312-5. doi: 10.1373/49.2.312. No abstract available. PMID 12560358
- [Background] Bonner RF, Emmert-Buck M, Cole K, Pohida T, Chuaqui R, Goldstein S, Liotta LA. Laser capture microdissection: molecular analysis of tissue. Science. 1997 Nov 21;278(5342):1481,1483. doi: 10.1126/science.278.5342.1481. No abstract available. PMID 9411767
- [Background] Emmert-Buck MR, Bonner RF, Smith PD, Chuaqui RF, Zhuang Z, Goldstein SR, Weiss RA, Liotta LA. Laser capture microdissection. Science. 1996 Nov 8;274(5289):998-1001. doi: 10.1126/science.274.5289.998. PMID 8875945
- [Background] Pease AC, Solas D, Sullivan EJ, Cronin MT, Holmes CP, Fodor SP. Light-generated oligonucleotide arrays for rapid DNA sequence analysis. Proc Natl Acad Sci U S A. 1994 May 24;91(11):5022-6. doi: 10.1073/pnas.91.11.5022. PMID 8197176
- [Background] Schena M, Shalon D, Davis RW, Brown PO. Quantitative monitoring of gene expression patterns with a complementary DNA microarray. Science. 1995 Oct 20;270(5235):467-70. doi: 10.1126/science.270.5235.467. PMID 7569999
- [Background] Sorlie T, Perou CM, Tibshirani R, Aas T, Geisler S, Johnsen H, Hastie T, Eisen MB, van de Rijn M, Jeffrey SS, Thorsen T, Quist H, Matese JC, Brown PO, Botstein D, Lonning PE, Borresen-Dale AL. Gene expression patterns of breast carcinomas distinguish tumor subclasses with clinical implications. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10869-74. doi: 10.1073/pnas.191367098. PMID 11553815
- [Background] Sgroi DC, Teng S, Robinson G, LeVangie R, Hudson JR Jr, Elkahloun AG. In vivo gene expression profile analysis of human breast cancer progression. Cancer Res. 1999 Nov 15;59(22):5656-61. PMID 10582678
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Ahr A, Holtrich U, Solbach C, Scharl A, Strebhardt K, Karn T, Kaufmann M. Molecular classification of breast cancer patients by gene expression profiling. J Pathol. 2001 Oct;195(3):312-20. doi: 10.1002/path.955. PMID 11673828
- [Background] Ahr A, Karn T, Solbach C, Seiter T, Strebhardt K, Holtrich U, Kaufmann M. Identification of high risk breast-cancer patients by gene expression profiling. Lancet. 2002 Jan 12;359(9301):131-2. doi: 10.1016/S0140-6736(02)07337-3. PMID 11809257
- [Background] West M, Blanchette C, Dressman H, Huang E, Ishida S, Spang R, Zuzan H, Olson JA Jr, Marks JR, Nevins JR. Predicting the clinical status of human breast cancer by using gene expression profiles. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11462-7. doi: 10.1073/pnas.201162998. Epub 2001 Sep 18. PMID 11562467
- [Background] Hedenfalk I, Duggan D, Chen Y, Radmacher M, Bittner M, Simon R, Meltzer P, Gusterson B, Esteller M, Kallioniemi OP, Wilfond B, Borg A, Trent J, Raffeld M, Yakhini Z, Ben-Dor A, Dougherty E, Kononen J, Bubendorf L, Fehrle W, Pittaluga S, Gruvberger S, Loman N, Johannsson O, Olsson H, Sauter G. Gene-expression profiles in hereditary breast cancer. N Engl J Med. 2001 Feb 22;344(8):539-48. doi: 10.1056/NEJM200102223440801. PMID 11207349
- [Background] Chicurel M. Faster, better, cheaper genotyping. Nature. 2001 Aug 9;412(6847):580-2. doi: 10.1038/35088146. No abstract available. PMID 11493890
- [Background] Hacia JG, Brody LC, Chee MS, Fodor SP, Collins FS. Detection of heterozygous mutations in BRCA1 using high density oligonucleotide arrays and two-colour fluorescence analysis. Nat Genet. 1996 Dec;14(4):441-7. doi: 10.1038/ng1296-441. PMID 8944024
- [Background] Hacia JG, Sun B, Hunt N, Edgemon K, Mosbrook D, Robbins C, Fodor SP, Tagle DA, Collins FS. Strategies for mutational analysis of the large multiexon ATM gene using high-density oligonucleotide arrays. Genome Res. 1998 Dec;8(12):1245-58. doi: 10.1101/gr.8.12.1245. PMID 9872980
- [Background] Staunton JE, Slonim DK, Coller HA, Tamayo P, Angelo MJ, Park J, Scherf U, Lee JK, Reinhold WO, Weinstein JN, Mesirov JP, Lander ES, Golub TR. Chemosensitivity prediction by transcriptional profiling. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10787-92. doi: 10.1073/pnas.191368598. PMID 11553813
- [Background] Alban A, David SO, Bjorkesten L, Andersson C, Sloge E, Lewis S, Currie I. A novel experimental design for comparative two-dimensional gel analysis: two-dimensional difference gel electrophoresis incorporating a pooled internal standard. Proteomics. 2003 Jan;3(1):36-44. doi: 10.1002/pmic.200390006. PMID 12548632
- [Background] Banks RE, Dunn MJ, Hochstrasser DF, Sanchez JC, Blackstock W, Pappin DJ, Selby PJ. Proteomics: new perspectives, new biomedical opportunities. Lancet. 2000 Nov 18;356(9243):1749-56. doi: 10.1016/S0140-6736(00)03214-1. PMID 11095271
- [Background] Adam PJ, Boyd R, Tyson KL, Fletcher GC, Stamps A, Hudson L, Poyser HR, Redpath N, Griffiths M, Steers G, Harris AL, Patel S, Berry J, Loader JA, Townsend RR, Daviet L, Legrain P, Parekh R, Terrett JA. Comprehensive proteomic analysis of breast cancer cell membranes reveals unique proteins with potential roles in clinical cancer. J Biol Chem. 2003 Feb 21;278(8):6482-9. doi: 10.1074/jbc.M210184200. Epub 2002 Dec 10. PMID 12477722
- [Background] Mikhitarian K, Reott S, Hoover L, Allen A, Cole DJ, Gillanders WE, Mitas M. Enhanced detection of RNA from paraffin-embedded tissue using a panel of truncated gene-specific primers for reverse transcription. Biotechniques. 2004 Mar;36(3):474-8. doi: 10.2144/04363RN01. No abstract available. PMID 15038162
- [Background] Mitas M, Mikhitarian K, Hoover L, Lockett MA, Kelley L, Hill A, Gillanders WE, Cole DJ. Prostate-Specific Ets (PSE) factor: a novel marker for detection of metastatic breast cancer in axillary lymph nodes. Br J Cancer. 2002 Mar 18;86(6):899-904. doi: 10.1038/sj.bjc.6600190. PMID 11953821
- [Background] Wallace MB, Block MI, Gillanders W, Ravenel J, Hoffman BJ, Reed CE, Fraig M, Cole D, Mitas M. Accurate molecular detection of non-small cell lung cancer metastases in mediastinal lymph nodes sampled by endoscopic ultrasound-guided needle aspiration. Chest. 2005 Feb;127(2):430-7. doi: 10.1378/chest.127.2.430. PMID 15705978
- [Background] Muller PY, Janovjak H, Miserez AR, Dobbie Z. Processing of gene expression data generated by quantitative real-time RT-PCR. Biotechniques. 2002 Jun;32(6):1372-4, 1376, 1378-9. PMID 12074169
- [Background] Mikhitarian, K., W.E. Gillanders, J.S. Almeida, R.H. Martin, J.C. Varela, J.S. Metcalf, D.J. Cole, and M. Mitas. 2005. Relative levels of gene expression are correlated with the ability to detect micrometastatic breast cancer: statistical analysis of data from a multi-institutional prospective cohort study and development of an innovative microarray strategy. Clin Cancer Res In Press.
- [Background] Mitas M, Almeida JS, Mikhitarian K, Gillanders WE, Lewin DN, Spyropoulos DD, Hoover L, Graham A, Glenn T, King P, Cole DJ, Hawes R, Reed CE, Hoffman BJ. Accurate discrimination of Barrett's esophagus and esophageal adenocarcinoma using a quantitative three-tiered algorithm and multimarker real-time reverse transcription-PCR. Clin Cancer Res. 2005 Mar 15;11(6):2205-14. doi: 10.1158/1078-0432.CCR-04-1091. PMID 15788668
- [Background] Mikhitarian K, Martin RH, Mitas M, Mauldin PD, Palesch Y, Metcalf JS, Cole DJ, Gillanders WE; Mims Study Group. Molecular analysis improves sensitivity of breast sentinel lymph node biopsy: results of a multi-institutional prospective cohort study. Surgery. 2005 Sep;138(3):474-81. doi: 10.1016/j.surg.2005.07.001. PMID 16213901
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu